CLINICAL TRIAL: NCT05321498
Title: A Phase 2, Randomized, Placebo-Controlled, Double-Blind Study of XPro1595 in Patients With Mild Cognitive Impairment (MCI) With Biomarkers of Inflammation
Brief Title: Study to Assess the Efficacy of XPro1595 in Patients With Mild Cognitive Impairment With Biomarkers of Inflammation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: MCI patients will now be enrolled in the XPro1595-AD-02 study.
Sponsor: Inmune Bio, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XPro1595-AD-03
Record Dates: First submitted 2022-03-03; First posted 2022-04-11 (Actual); Last update posted 2023-09-28 (Actual); Status verified 2023-09

CONDITIONS: Mild Cognitive Impairment (MCI); Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders
Keywords: Inflammation; Biomarker; Tumor Necrosis Factor (TNF)
MeSH Terms: conditions — Cognitive Dysfunction; Alzheimer Disease; Dementia; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Tauopathies; Neurodegenerative Diseases; Mental Disorders; Inflammation | interventions — XENP 1595

STUDY DESIGN:
Intervention Model Description: * (2:1) XPro1595 (1mg/kg), placebo
  * Weekly subcutaneous injections
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 1.0 mg/kg XPro1595 (Experimental): 1.0 mg/kg XPro1595 will be administered via subcutaneous injection once a week for 12 weeks.
  Interventions: Drug: XPro1595
- 1.0 mg/kg Placebo (Placebo Comparator): 1.0 mg/kg of Placebo will be administered via subcutaneous injection once a week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: XPro1595 — XPro1595 will be delivered by subcutaneous injection once a week.
  Other Names: INB03/XPro™; XENP1595; Dominant-negative Tumor Necrosis Factor (DN-TNF)
  Arms: 1.0 mg/kg XPro1595
Drug: Placebo — Placebo will be delivered by subcutaneous injection once a week
  Other Names: Matching Placebo
  Arms: 1.0 mg/kg Placebo

SUMMARY:
The goal of this Phase 2 MCI study is to determine whether 1.0 mg/kg XPro1595 is superior to placebo at improving measures of cognition, functioning and brain quality in individuals with MCI and biomarkers associated with neuroinflammation (APOE4) and to evaluate safety, tolerability, and efficacy of XPro1595.

DETAILED DESCRIPTION:
This study is designed as a Phase 2, double-blind randomized, placebo-controlled study investigating the safety, tolerability, and efficacy of XPro1595 in patients with MCI. The planned dose is 1.0 mg/kg of XPro1595 and matching placebo.

ELIGIBILITY:
Inclusion Criteria:

Patients are eligible to be included in the study only if all the following criteria apply:

* Adult male and female patients ≥ 55 years to ≤ 80 years of age at the time of consent;
* Diagnosed with MCI of probable Alzheimer's disease (Albert 2011; National Institute on Aging - Alzheimer's Association [NIA-AA]). Patients who have received previous therapy for Alzheimer's disease may still be eligible;
* Amyloid positive (documented in medical history or assessed during screening through blood test);
* Literate and capable of reading, writing, and communicating effectively with others, based on the PI's assessment;
* Has a study partner willing to participate for the duration of the trial who either lives in the same household or interacts with the patient at least 4 hours per day and on at least 4 days per week, who is knowledgeable about the patient's daytime and night-time behaviors and who can be available to attend all clinic visits in person at which informant assessments are performed.

Exclusion Criteria:

* Have any contraindications to MRI scanning, including cardiac pacemaker/defibrillator, ferromagnetic metal implants (e.g., in-skull and cardiac devices other than those approved as safe for use in MRI scanners at the strength required for this study);
* Receives considerable help to carry out basic ADL living either in the home or as a resident in a nursing home or similar facility;
* Lifetime history of a major psychiatric disorder including schizophrenia and bipolar disorder. Major depressive disorder that has resulted in 2 or more hospitalizations in a lifetime. Major depressive episode during the past 5 years that is judged by the clinical team unlikely to have been part of Alzheimer's prodrome. History of suicidality: has answered "yes" to Columbia-Suicide Severity Rating Scale (C-SSRS) suicidal ideation items 4 or 5, or any suicidal behavior within 6 months before Screening, at Screening, or at the Week 1 Visit, or has been hospitalized or treated for suicidal behavior in the past 5 years before Screening;
* History of substance abuse within 12 months; use of cannabis or cannabis products within 6 months of consent;
* Enrolled in another clinical trial where patients receive treatment with an investigational drug or treatment device or have received treatment on another AD clinical trial within the last 60 days from Day 1

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-06 (Estimated); Primary Completion 2023-10-26 (Estimated); Study Completion 2023-10-26 (Estimated)

PRIMARY OUTCOMES:
Change in Early and Mild Alzheimer's Cognitive Composite (EMACC) | 12 Weeks
  Change from Baseline to Week 12 in the Early and Mild Alzheimer's Cognitive Composite (EMACC) (Jaeger 2017) made up of the following tests:
  * International Shopping List Test- Immediate recall (Word List Learning Test-Immediate recall)
  * Trail Making Test Part A and B
  * Digit Symbol Coding Test
  * Digit Span Forward and Backward
  * Category Fluency Test (DKEFS)
  * Letter Fluency Test (DKEFS)
  To assess the efficacy of XPro1595 compared with placebo on cognitive performance in patients with MCI

SECONDARY OUTCOMES:
Change in Mean Computer-based Cognitive Assessment (Cogstate) Composite score from Screening to Week 12 | 12 Weeks
  Change from Screening to Week 12 in Cogstate Composite mean score.
  Cogstate is a brief, computerized, neuropsychological battery to evaluate cognitive impairments in mild cognitive impairment (MCI), and Alzheimer's disease (AD). CogState assesses attention and memory functions - including Information processing speed, Visual attention, Working memory and Visual learning. Cogstate scores are measured on a linear scale (with no maximum score). A reduction in scores compared to baseline signifies an improvement in cognitive functions.
  The Cogstate battery will be administered at Screening and each week for 12 weeks.
  To assess the efficacy of XPro1595 compared with placebo on cognitive performance in patients with MCI
Change in myelin content | 12 Weeks
  Change from Screening to Week 12 in myelin content.
Change in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker amyloid) | 12 Weeks
  Change from Screening to Week 12 in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker amyloid)
  To assess the efficacy of XPro1595 compared with placebo on blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker amyloid)
Change in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau) | 12 Weeks
  Change from Screening to Week 12 in blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau)
  To assess the efficacy of XPro1595 compared with placebo on blood inflammatory and neurodegeneration biomarkers (on blood inflammatory and neurodegeneration biomarker pTau)
Change in Imaging (MRI) Neuroinflammation | 12 Weeks
  Change from Screening to Week 12 in MRI neuroinflammation (White matter Free Water)
  To assess the efficacy of XPro1595 compared with placebo on imaging neuroinflammation
Change in imaging markers of brain quality | 12 Weeks
  Change from Screening to Week 12 in regional brain glucose uptake as measured by F-fluorodeoxyglucose-Positron Emission Tomography (FDG-PET) scans
  Alzheimer's Disease (AD) is characterized by a chronic brain glucose deficit. White matter glucose deterioration is also evident in Mild Cognitive Impairment (MCI) and specific to limbic fascicles. We will quantify the change in regional brain glucose uptake for gray matter and white matter tracts using PET imaging and the F-fluorodeoxyglucose (FDG) radiotracer. PET maps will be registered to Magnetic Resonance (MR) anatomical images and corrected for partial volume effect. Standard uptake value ratios (SUVr) will be calculated using the cerebellum as a reference region.
  FDG-PET scans will be performed at Screening and Week 12.
  To assess the efficacy of XPro1595 compared with placebo on imaging markers of brain quality
Change in apparent fiber density (AFD) | 12 Weeks
  Change from Baseline to Week 12 in MRI Apparent Fiber Density (AFD)
  To assess the efficacy of XPro1595 compared with placebo on axonal integrity in patients with MCI
Change in non-cognitive behavioral symptoms | 12 Weeks
  Change from Screening to Week 12 in Neuropsychiatric Inventory (NPI-12) study partner items
  To assess the effect of XPro1595 compared with placebo on non-cognitive behavioral symptoms in patients with MCI
Change in brain activity | 12 Weeks
  Change from Screening to Week 12 in brain activity as measured by electroencephalogram (EEG) scans (Change in brain activity as measured by the EEG in microvolts).
  Specifically, a series of EEG markers previously associated with AD (Horvath et al. 2018) including high and low frequency band powers, the P300, and Mismatch Negativity (MMN) event-related potentials will be evaluated.
  An EEG scan will be administered at Screening and each week for 12 weeks.
  To assess the efficacy of XPro1595 compared with placebo on brain activity in patients with MCI
Change in speech and language | 12 Weeks
  Change from Baseline to Week 12 in language and speech patterns using Winterlight Labs analysis
  To assess the effect of XPro1595 compared with placebo on speech and language in patients with MCI
Change in Alzheimer's Disease Cooperative Study - Mild Cognitive Impairment Activities of Daily Living (ADCS-MCI ADL) | 12 Weeks
  Change from Screening to Week 12 in Alzheimer's Disease Cooperative Study - Mild Cognitive Impairment Activities of Daily Living (ADCS-MCI ADL)
  The 23-item ADCS-MCI-ADL Scale has good test-retest reliability, will be utilized to assess performance functioning in MCI patients (Galasko et al., 1997; Douglas Galasko et al., 2006; Pedrosa et al., 2010). The ADCS-ADL includes 18 items from traditional basic ADL scales and 5 items from instrumental activities of daily living scales (IADL) The possible range of total scores for the ADL Scale is 0-53 and higher scores indicate better functioning. The internal reliability was .91( Galasko et al., 1997; Douglas Galasko et al., 2006; Pedrosa et al., 2010).
  The ADCS-MCI ADL will be performed at Screening and Week 12.
  To assess the effect of XPro1595 compared with placebo on Activities of Daily Living (ADL) in patients with MCI
Change in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) | 12 Weeks
  Change from Screening to Week 12 in Clinical Dementia Rating Scale Sum of Boxes (CDR-SB)
  The CDR scale is a clinician-rated dementia staging system that tracks the progression of cognitive impairment in 6 categories (memory, orientation, judgement and problem solving, community affairs, home and hobbies, and personal care). Each category is scored on a 5-point scale in which None = 0, Questionable = 0.5, Mild = 1, Moderate = 2, and Severe = 3. The global CDR score is established by clinical scoring rules and has values of 0 (no dementia), 0.5, (questionable dementia), 1 (mild dementia), 2 (moderate dementia), and 3 (severe dementia). The Clinical Dementia Rating Scale Sum of Boxes (CDR-SB) is obtained by adding the ratings in each of the 6 categories and ranges from 0 to 18 with higher scores indicative of greater impairment.
  To assess the effect of XPro1595 compared with placebo on cognition and global function in patients with MCI
Number of participants who experience adverse events and serious adverse events | Screening up to 28 days post last dose
  Clinically significant abnormalities of laboratory values, physical findings, electrocardiogram findings and other safety assessments will be recorded as adverse events if the findings meet the defined criteria for adverse events.

OTHER OUTCOMES:
Change in Goal Attainment Scale (GAS) | 12 Weeks
  Change in Goal Attainment Scale (GAS)
  The achievement of each goal is rated on a 5-point attainment scale (-2, -1, 0, +1, +2) to allow standardized scoring of personalized outcomes. A participant's overall goal attainment is quantified using a formula that takes into account the number of goals that have been set, and the extent to which they are correlated with each other. For each identified goal area, the caregiver will be asked to give a detailed description of the patient's current (baseline) status and goal status, which will be recorded at the -1 and 0 levels on the 5-point scale, respectively. The remaining levels of the scale will then be set: somewhat better than the goal (+1), much better than the goal (+2), and much worse than the goal (-2).
  To evaluate the effect of XPro1595 compared with placebo on goal attainment scores
Change in measures of activity | 12 Weeks
  Change from Screening to Week 12 in activity metrics (time spent lying, sitting, standing, stepping, upright, in walking bouts, in-context specific walking bouts; number of steps, and sit-to-stand transitions) as measured by the activity monitor. Physical activity will be measured in real time using the activity monitor worn on the patient's wrist. Total activity counts per minute (higher activity counts = more activity) and number of steps taken will be derived from data. Patients will be equipped with the monitoring device during the screening period and activity metrics will be measured for 7 days prior to each EMACC assessment. Data will be measured at Screening, Week 1, Week 3, Week 6, Week 9 and Week 12.
  To assess the effect of XPro1595 compared to placebo on measures of activity
Evaluate predictability of patient response after placebo administration and potential influence of study partners on outcome evaluation using the Multidimensional Psychological Questionnaire (MPsQ) with a 5 point scale | 12 Weeks
  The Multidimensional Psychological Questionnaire (MPsQ) questionnaires have been designed to specifically measure patient personality characteristics associated with the placebo response. The MPsQ questionnaires are self-reported, and each item is rated on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree).
  MPsQs will be completed by the patient and separate MPsQs will be completed by the study partner at screening.
  MPsQs will be completed by the patient and separate MPsQs will be completed by the study partner prior to investigational product administration.
  The patient and study partner will complete MPsQs at Screening and Week 1.
  To measure patient personality characteristics associated with the placebo response.

CONTACTS AND LOCATIONS:
Overall Officials: Tara Lehner, Study Director — INmune Bio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Alvarez A, Cacabelos R, Sanpedro C, Garcia-Fantini M, Aleixandre M. Serum TNF-alpha levels are increased and correlate negatively with free IGF-I in Alzheimer disease. Neurobiol Aging. 2007 Apr;28(4):533-6. doi: 10.1016/j.neurobiolaging.2006.02.012. Epub 2006 Mar 29. PMID 16569464
- [Background] Bongartz T, Sutton AJ, Sweeting MJ, Buchan I, Matteson EL, Montori V. Anti-TNF antibody therapy in rheumatoid arthritis and the risk of serious infections and malignancies: systematic review and meta-analysis of rare harmful effects in randomized controlled trials. JAMA. 2006 May 17;295(19):2275-85. doi: 10.1001/jama.295.19.2275. PMID 16705109
- [Background] Buchhave P, Zetterberg H, Blennow K, Minthon L, Janciauskiene S, Hansson O. Soluble TNF receptors are associated with Abeta metabolism and conversion to dementia in subjects with mild cognitive impairment. Neurobiol Aging. 2010 Nov;31(11):1877-84. doi: 10.1016/j.neurobiolaging.2008.10.012. Epub 2008 Dec 13. PMID 19070941
- [Background] Chance SA, Clover L, Cousijn H, Currah L, Pettingill R, Esiri MM. Microanatomical correlates of cognitive ability and decline: normal ageing, MCI, and Alzheimer's disease. Cereb Cortex. 2011 Aug;21(8):1870-8. doi: 10.1093/cercor/bhq264. Epub 2011 Jan 14. PMID 21239393
- See also: Alzheimer's Association annual report releasing statistics regarding Alzheimer's disease — https://www.alz.org/alzheimers-dementia/facts-figures